CLINICAL TRIAL: NCT07122258
Title: To Investigate the Safety of the CAROL Device for Lung Tumour Treatment in Patients With Non-small Cell Lung Cancer Tumours(s) ≤ 2 cm (cT1b)
Brief Title: Early Feasibility Study (EFS) of the 'CAROL' for Treatment of Lung Cancer Stage 1
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tau Medical Australia Pty Ltd (Industry)
Collaborators: Tau-MEDICAL Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Tau-MEDICAL Co., Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAROL
Record Dates: First submitted 2025-07-20; First posted 2025-08-14 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: NSCLC (Non-small Cell Lung Cancer)
Keywords: CAROL; TAU MEDICAL
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Intervention Model Description: Multi-center, open label, single arm, early feasibility study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAROL Device Treatment for Early-Stage NSCLC (Experimental): Participants in this single-arm study will undergo treatment with the CAROL device for localized lung tumors (NSCLC ≤ 2 cm, cT1b). All participants will receive a single CAROL procedure using a conformable electrode, followed by surgical resection of the tumor.
  The first 3 sentinel participants will receive a maximum dose of 0.3 mL of the conformable electrode. The next 4 participants will receive up to 2.0 mL. Safety and preliminary efficacy will be assessed through scheduled follow-up visits, including imaging, pulmonary function testing, laboratory assessments and pain monitoring.
  Adverse events will be monitored throughout the study, with grading based on CTCAE v5.0, specifically focusing on "Respiratory, thoracic, and mediastinal disorders." The study includes visits at screening, pre-procedure, post-procedure (24-36 hours), pre- and post-resection, and follow-up at approximately one and three months.
  Interventions: Device: CAROL NSCLC treatment Device

INTERVENTIONS:
Device: CAROL NSCLC treatment Device — Participants in this single-arm study will undergo treatment with the CAROL device for localized lung tumors (NSCLC ≤ 2 cm, cT1b). All participants will receive a single CAROL procedure using a conformable electrode, followed by surgical resection of the tumor.
  The first 3 sentinel participants will receive a maximum dose of 0.3 mL of the conformable electrode. The next 4 participants will receive up to 2.0 mL. Safety and preliminary efficacy will be assessed through scheduled follow-up visits, including imaging, pulmonary function testing, laboratory assessments and pain monitoring.
  Adverse events will be monitored throughout the study, with grading based on CTCAE v5.0, specifically focusing on "Respiratory, thoracic, and mediastinal disorders." The study includes visits at screening, pre-procedure, post-procedure (24-36 hours), pre- and post-resection, and follow-up at approximately one and three months.

SUMMARY:
This study aims to evaluate the safety of the CAROL device for treating lung tumors in patients diagnosed with non-small cell lung cancer (NSCLC) with tumor size ≤ 2 cm (cT1b). The primary objective is to assess safety by monitoring and grading adverse events using the CTCAE v5.0 criteria at one month following the procedure.

ELIGIBILITY:
Inclusion Criteria:

Those who meet all the following criteria are eligible to participate in the clinical trial.

1. Adults 18 years of age or older at the time of screening
2. NSCLC tumour(s)≤ 2 cm (cT1b) suitable for resection
3. Suitable candidate for resection per standard of practice (Lobectomy)
4. NSCLC is confirmed pathologically for the tissue that will be ablated
5. Location of tumour:

   * ① in outer one thirds of lung (between outermost 1/3 measured by tumour centre),
   * ② if the centre of the tumour is located within the outermost 1/3, inclusion will proceed,
   * ③ anticipation that resection (lobectomy) would remove all gross tumour and ablation with grossly negative margins,
   * ④ one or more radiofrequency ablation (RFA) applications would target entire margin according to the RFA plan
6. Signed free and informed consent as prescribed by hospital policies.

Exclusion Criteria:

Those who meet any of the following criteria are excluded from this clinical trial.

1. Centralised tumour (inner most one third) not amenable to resection (abutting main stem bronchus, main pulmonary artery branches, oesophagus or trachea)
2. Other primary lung tumours
3. Tumour is associated with vulnerable zone of pleural effusion
4. If the centre of the tumour is not located within the outermost 1/3, exclusion will proceed
5. PFT: post-bronchodilator forced expired volume in on second (FEV1) or forced vital capacity (FVC) ≤60% predicted, diffusing capacity of the lung for carbon monoxide (DLCO) ≤ 50% predicted
6. Patients with evidence of severe chronic pulmonary disease including asthma, Chronic Obstructive Pulmonary Disease (COPD), or Interstitial Lung Disease (ILD).
7. Requirement of supplemental oxygen at rest or exercise
8. Hospitalization for cardiac disease within the preceding 3 months
9. Liver enzymes (Alanine Aminotransferase [ALT], Alkaline Phosphatase [ALP], Aspartate Aminotransferase [AST]) or total bilirubin >1.5 upper limit of normal (ULN)
10. Serum creatinine > 2 mg/dl
11. Recent infection (within 30 days)
12. Receiving immunosuppressive medication or prednisone > 20 mg/day (or equivalent)
13. Pre-existing implants - either within the airways or any other location - that impede navigation to or visualisation of the target lesion, in the opinion of the investigator
14. Pregnant or breastfeeding women and those of childbearing potential who are not practicing a reliable form of contraception.
15. Disorder of coagulation, history of severe haemoptysis, or receiving anticoagulant medication. Antiplatelet medication is permitted provided that the medication can be held a minimum of 7 days prior to the procedures and 10 days post-procedures, where this refers to both the ablation and surgical procedures
16. Any condition or anatomical factor that, in the opinion of the investigator or reviewer, may interfere with the safety of the patient, the conduct of the procedure, or evaluation of the study objectives (e.g. severe bronchial narrowing, wall compromise)
17. Any tumour characteristic that in the opinion of the investigator or reviewers may interfere with the safety of the patient or evaluation of the study objectives
18. Contraindication to complete neuromuscular blockade during the ablation procedure
19. Implantable cardiac devices such as pacemakers or defibrillators, especially with unipolar electrode configurations
20. Known hypersensitivity or allergy to gallium, indium, or other components of the conformable electrode
21. Medically inoperable conditions
22. Participant who is currently participating in, or planning to participate in (during the course of the trial), another non-observational clinical research study
23. Participants who have participated in a non-observational clinical research study within either the past 30 days or who are still within the intervention's wash-out period (whichever is longer)
24. Participant who, in the opinion of the investigator, is not suitable for participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Common Terminology Criteria for Adverse Events(CTCAE) | 1 month post-procedure
  Graded using CTCAE grade (v5.0) criteria(CTCAE) The CTCAE utilizes a scale ranging from Grade 1 (mild) to Grade 5 (death-related) to classify the severity of adverse events. A higher CTCAE grade indicates increased severity of the adverse event, signifying a worse outcome.

SECONDARY OUTCOMES:
Device success | Immediately after application (measured by imaging during the procedure)
  Success rate of CAROL device positioning at the target site The success rate of CAROL device positioning at the target site immediately after application, as assessed by fluoroscopic imaging and /or bronchoscopic visualization during the procedure. Proper positioning is defined as complete coverage of the target segmental bronchus by the ablation electrode without malposition or dislodgement. Frequencies and percentages will be presented to summarise the success rate.
Procedural success | Immediately after procedure (intraoperative and early postoperative period)
  Successful delivery of the ablation treatment for lung cancer using the CAROL system, performed according to the Instruction for Use (IFU) and treatment plan. Success will be determined based on the following criteria:
  Successful delivery of the CAROL catheter to the target site Successful injection of the Conformable Electrode (E-GaIn) Achievement of target ablation temperature Retrieval of the device without malfunction
Procedural success | 5 ~ 10 days after lung resection
  Pathological analysis Pathological evidence of effective ablation will be evaluated using hematoxylin and eosin (H&E) staining to assess tissue viability. The extent of the coagulative necrotic zone relative to the tumor location will be quantified by pathologists. Descriptive statistics (mean, range) will summarize the extent of ablation effectiveness.
Procedural success | 2~9 days after the CAROL procedure
  Imaging data evaluation Imaging data from computed tomography (CT) scans will be assessed to evaluate the extent of ablation, including lesion size and ablation margin relative to baseline. Measurements will be reviewed by radiologists using standard radiologic assessment criteria. Descriptive statistics will be presented for changes in treated areas.

OTHER OUTCOMES:
Evaluation of Quality of Life scores | 2~9 days after CAROL the procedure
  Evaluation of Quality of Life scores(EQ-5D) The EQ-5D questionnaire will be used to assess patient's health-related quality of life. The EQ-5D includes 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression), each scored on 5 levels.
  Scores will be converted to an index value ranging from -0.594 (worst health state) to 1.000 (perfect health), based on country-specific value sets. Higher scores indicate better health-related quality of life.
Evaluation of pain scores | 2~9 days after the CAROL procedure
  Visual Analogue Scale (VAS) Pain intensity will be assessed using the Visual Analogue Scale (VAS), a validated instrument consisting of a 10 cm horizontal line anchored by "no pain" (0) and "worst imaginable pain" (10). Participants will be asked to indicate their current level of pain on the scale. Higher scores indicate greater pain severity.
Predicted and actual volume of liquid metal delivered | 6~14 days after the CAROL procedure
  The volume of Conformable Electrode (E-GaIn) predicted during the planning phase will be compared with the actual volume delivered during the CAROL procedure. Measurements will be obtained from procedure records and delivery system readouts. Differences will be quantified in milliliters (mL) and summarized using descriptive statistics.
Predicted and actual ablation size | 6 to 14 days after the CAROL procedure
  The ablation size predicted during pre-treatment planning will be compared to the actual ablation zone measured by post-procedural imaging. Ablation volume will be quantified in cubic centimeters (cm3) using CT or MRI data, and descriptive statistics will be used to summarize differences.
Distribution pattern of conformable electrode in varying bronchial anatomies | Day 23 to Day 37 after the CAROL procedure
  CT images will be used to assess the spatial distribution of the Conformable Electrode (E-GaIn) across different bronchial structures. Anatomical coverage (e.g., lobar/segmental bronchi), symmetry, and dispersion pattern will be visually classified and quantitatively measured by independent radiologists. Descriptive statistics will summarize the observed distribution patterns.
Feasibility of procedural planning in various bronchial geometries | Day 23 to Day 37 after the CAROL procedure
  The feasibility of procedural planning will be assessed based on whether the planned delivery paths through bronchial geometries were technically achievable during procedure simulation using CT-based airway mapping.
Accuracy of procedural planning in various bronchial geometries | Day 23 to Day 37 after the CAROL procedure
  Accuracy will be assessed by comparing the planned device path (based on CT-based bronchial mapping) with the actual path and final position as observed in post-procedure CT imaging. The deviation between the planned and actual paths will be measured in millimeters in three-dimensional space by independent radiologists. Descriptive statistics (mean, standard deviation, and range) will be used to summarize the accuracy for each bronchial geometry type (e.g., lobar, segmental).
User feedback score on device usability and operating handling characteristics | Day 23 to Day 37 after the CAROL procedure
  User feedback will be collected using a standardized questionnaire assessing device usability and operating handling characteristics, including perceived ease of use, catheter maneuverability, and procedural confidence. Responses will be summarized using descriptive analysis of response frequencies and thematic grouping of any free-text comments.